CLINICAL TRIAL: NCT03997019
Title: Ultrasound Guided Erector Spinae Plane Block in Cardiac Surgery
Brief Title: Erector Spinae Plane Block in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FXLD
Record Dates: First submitted 2019-02-20; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: group A WILL RECEIVE OPOID analgesia group B will receive ESP block
Who Masked: Participant, Outcomes Assessor
Masking Description: both patient and data collector will be unaware of the group nature
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): opioid analgesia
  Interventions: Procedure: opioid analgesia
- group B (Active Comparator): ESP block
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: opioid analgesia — opioid analgesia will be used with general anaesthesia
  Arms: group A
Procedure: ESP block — ultrasound guided ESP Block before anaesthesia induction
  Arms: group B

SUMMARY:
ultrasound guided bilateral erector spinae plane block will be used as adjuvant to general anaesthesia in cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* elective surgery

Exclusion Criteria:

* emergency
* patient refusal
* infection at or near catheter insertion

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
pain score | 48 hours
  NRS will be used to assess pain

SECONDARY OUTCOMES:
anaesthesia consumption | 6 hours
  cumulative anaesthesia MAC
ultrasound guided postoperative diaphragmatic excursion | 24 hours
  diaphragmatic movement during inspiration an expiration
spirometric respiratory funtion | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No